CLINICAL TRIAL: NCT06719219
Title: A Phase I, Randomized, Double-Blinded and Controlled Trial to Evaluate Safety and Immunogenicity of an Investigational Multicomponent Staphylococcus Aureus Toxoid Vaccine (LTB-SA7) in Healthy Adults.
Brief Title: A First in Human Trial to Assess the Safety and Immunogenicity of LTB-SA7 Vaccine Against Staphylococcus Aureus.
Acronym: LTBSA701
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LimmaTech Biologics AG (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other); Navy Medical Research Command (NMRC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LTBSA701; 75A50122C00028 (Other Grant/Funding Number: Health and Human Services and Biomedical Advanced Research and Development Authority); WT224842 (Other Grant/Funding Number: Wellcome Trust); Agmt dtd 2/28/2023 (Other Grant/Funding Number: UK Department of Health and Social Care as part of the Global Antimicrobial Resistance Innovation Fund); Agmt dtd 1/30/2023 (Other Grant/Funding Number: Germany's Federal Ministry of Education and Research)
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Staphylococcus (S.) Aureus Infection
Keywords: Staphylococcus aureus vaccine; skin and soft tissue infection vaccine; staphylococcus aureus recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- LTB-SA7 low dose, 1 vaccination (Experimental): The candidate toxoid vaccine (LTB-SA7) is administered once, 1 month later participant receives a placebo.
  Interventions: Biological: LTB-SA7
- LTB-SA7 low dose, 2 vaccinations (Experimental): The candidate toxoid vaccine (LTB-SA7) is administered twice, 1 month apart.
  Interventions: Biological: LTB-SA7
- LTB-SA7 medium dose, 1 vaccination (Experimental): The candidate toxoid vaccine (LTB-SA7) is administered once, 1 month later participant receives a placebo.
  Interventions: Biological: LTB-SA7
- LTB-SA7 medium dose, 2 vaccinations (Experimental): The candidate toxoid vaccine (LTB-SA7) is administered twice, 1 month apart.
  Interventions: Biological: LTB-SA7
- LTB-SA7 high dose, 1 vaccination (Experimental): The candidate toxoid vaccine (LTB-SA7) is administered once, 1 month later participant receives a placebo.
  Interventions: Biological: LTB-SA7
- LTB-SA7 high dose, 2 vaccinations (Experimental): The candidate toxoid vaccine (LTB-SA7) is administered twice, 1 month apart.
  Interventions: Biological: LTB-SA7
- Placebo (Placebo Comparator): Participant receives placebo twice, 1 month apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LTB-SA7 — LTB-SA7 is a toxoid based vaccine consisting of five components including seven toxoids formulated with Alhydrogel.
  Arms: LTB-SA7 high dose, 1 vaccination; LTB-SA7 high dose, 2 vaccinations; LTB-SA7 low dose, 1 vaccination; LTB-SA7 low dose, 2 vaccinations; LTB-SA7 medium dose, 1 vaccination; LTB-SA7 medium dose, 2 vaccinations
Biological: Placebo — Sodium Phosphate with Sodium Chloride
  Arms: Placebo

SUMMARY:
In this study, the candidate vaccine LTB-SA7 will be tested for safety and immunogenicity in healthy adults.

DETAILED DESCRIPTION:
LTB-SA7 is a candidate vaccine designed to induce immune response against toxins produced by Staphylococcus aureus. During the study, healthy adults will be randomized to receive one out of three different vaccine doses (starting with the group receiving the lowest dose), or a placebo. Participants will receive 2 injections, either two with candidate vaccine, 1 vaccine and 1 placebo, or 2 times placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health by medical history, laboratory findings and physical examination as judged by the investigator before receiving the first injection.
2. Participant who is willing and able to comply with the requirements of the protocol (e.g., completion of the diary forms, return for follow-up visits).
3. Signed written informed consent obtained from the participant.
4. Participants between 18-50 years (inclusive) of age at the time of the first injection.
5. Negative urine pregnancy test for women of childbearing potential (WOCBP).
6. WOCBP must be willing to use a highly effective method of contraception during the trial.

Exclusion Criteria:

1. Health conditions that, in the opinion of the investigator, may interfere with optimal participation in the trial or place the participant at increased risk of adverse events.
2. Any deviation from the normal range in biochemistry or hematology blood tests clinically significant in the opinion of the investigator, measured at the screening visit.
3. Clinically significant abnormalities on physical examination.
4. Suspected or known hypersensitivity (including allergy) to any of the vaccine components or medical equipment whose use is foreseen in this trial.
5. History of allergy to any vaccine.
6. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws (e.g., coagulation disorder).
7. Known or suspected impairment of immunological function e.g., documented Human Immunodeficiency Virus (HIV) infection, asplenia/splenectomy, or history of autoimmune disease or lymphoproliferative disorder.
8. Positive blood test for HBsAg, HCV, HIV-1/2.
9. History of systemic administration of immunosuppressive drugs, i.e., corticosteroids, (PO/IV/IM) within the last month prior to vaccination or for more than 14 consecutive days within 3 months prior to vaccination, until the last blood sampling visit (i.e., prednisone or equivalent ≥20 mg/day). Inhaled and topical steroids are allowed.
10. Administration of antineoplastic and immune-modulating agents or chemotherapy within 3 months prior to vaccination.
11. Planned or actual administration of any licensed vaccine within 14 days prior to each vaccination and 30 days after each vaccination. Note: In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organized by the public health authorities, the time period described above can be reduced, if necessary, for that vaccine provided it is licensed or authorized and used according to the local governmental recommendations and provided a written approval of the Sponsor is obtained.
12. Concurrently participating in another clinical trial, at any time during the trial period, in which the participant has been or will be exposed to an investigational or a non-investigational interventional vaccine/ product (pharmaceutical product).
13. Body Mass Index (BMI) ≤19 or ≥35
14. History of any chronic or progressive disease that according to judgment of the investigator could interfere with the trial outcomes or pose a threat to the participant's health.
15. Received an investigational or non-registered product (medicinal drug or vaccine), other than the trial vaccine within 3 months prior to 1st administration of trial vaccine, or planned use during the trial period.
16. Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of trial vaccine.
17. Blood donation equal or greater to 500 mL of blood drawn within 3 months preceding the first or second vaccination or planned during the trial period as reported by the participant.
18. Use of any systemic antibiotic therapy within 1 week preceding each vaccination.
19. Participants with an elective surgical intervention, planned during the trial period until 1 month after 2nd vaccination.
20. Female participants lactating, pregnant, or intending to become pregnant as reported by the participant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety - Solicited local and systemic AEs | During 7 days following each vaccination.
  Occurrence and severity of solicited local and systemic AEs during 7 days after each dose (i.e., day of vaccination and the 6 subsequent days) in all participants by intervention group.
Safety - Unsolicited AEs | During 28 days following each vaccination.
  Occurrence, severity, and relationship to vaccination of unsolicited AEs during 28 days after each dose (i.e., day of injection and the 27 subsequent days) in all participants by intervention group.
Safety - SAEs | Throughout the study, on average 8 months
  Occurrence, severity, and relationship to vaccination of SAEs in all participants during the trial duration by intervention group.
Immunogenicity - GMTs of anti-toxoids IgGs in serum at V4 | 1 month from the first vaccination.
  Serum IgG antibody geometric mean titers (GMT) against each of the 7 toxoids present in the LTB-SA7 vaccine in serum samples collected 4 weeks after the 1st vaccination (Visit 4 [Day 29]) by intervention group to identify preferred dose(s).

SECONDARY OUTCOMES:
Immunogenicity - GMTs of anti-toxoid IgGs in serum at V3, V5 and V6 | From 1 week after first vaccination till Day 57 (Visit 6).
  Serum IgG antibody geometric mean titers (GMT) against each of the 7 toxoids present in the LTB-SA7 vaccine in samples collected 1 week after 1st and 2nd vaccination and 4 weeks after 1st and 2nd vaccination (Visit 3 [Day 8], Visit 5 [Day 36], and Visit 6 [Day 57]).
Immunogenicity - GMFR of anti-toxoid IgGs in serum at V2-V6. | Between baseline on Visit 2 (Day 1) until 4 weeks post 2nd vaccination on Visit 6 (Day 57).
  Serum IgG antibody geometric mean fold ratio (GMFR) vs. baseline.
Immunogenicity - Total IgGs titer in serum | Between baseline on Visit 2 (Day 1) until 4 weeks post 2nd vaccination on Visit 6 (Day 57).
  Percentage of participants with ≥ 2-fold ≥ 4-fold, and ≥ 8-fold IgG titer increase vs. baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nehkonti Adams, MD, Principal Investigator — Naval Medical Research Command
Locations (1):
- Naval Medical Research Command Clinical Trial Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoergenhofer C, Gelbenegger G, Hasanacevic D, Schoner L, Steiner MM, Firbas C, Buchtele N, Derhaschnig U, Tanzmann A, Model N, Larcher-Senn J, Drost M, Eibl MM, Roetzer A, Jilma B. A randomized, double-blind study on the safety and immunogenicity of rTSST-1 variant vaccine: phase 2 results. EClinicalMedicine. 2024 Jan 5;67:102404. doi: 10.1016/j.eclinm.2023.102404. eCollection 2024 Jan. PMID 38274114
- [Background] Rajagopalan G, Iijima K, Singh M, Kita H, Patel R, David CS. Intranasal exposure to bacterial superantigens induces airway inflammation in HLA class II transgenic mice. Infect Immun. 2006 Feb;74(2):1284-96. doi: 10.1128/IAI.74.2.1284-1296.2006. PMID 16428778
- [Background] Nizet V. Understanding how leading bacterial pathogens subvert innate immunity to reveal novel therapeutic targets. J Allergy Clin Immunol. 2007 Jul;120(1):13-22. doi: 10.1016/j.jaci.2007.06.005. PMID 17606031
- [Background] Tattevin P, Schwartz BS, Graber CJ, Volinski J, Bhukhen A, Bhukhen A, Mai TT, Vo NH, Dang DN, Phan TH, Basuino L, Perdreau-Remington F, Chambers HF, Diep BA. Concurrent epidemics of skin and soft tissue infection and bloodstream infection due to community-associated methicillin-resistant Staphylococcus aureus. Clin Infect Dis. 2012 Sep;55(6):781-8. doi: 10.1093/cid/cis527. Epub 2012 Jun 5. PMID 22670044
- [Background] Tong SY, Davis JS, Eichenberger E, Holland TL, Fowler VG Jr. Staphylococcus aureus infections: epidemiology, pathophysiology, clinical manifestations, and management. Clin Microbiol Rev. 2015 Jul;28(3):603-61. doi: 10.1128/CMR.00134-14. PMID 26016486
- [Background] Tran VG, Venkatasubramaniam A, Adhikari RP, Krishnan S, Wang X, Le VTM, Le HN, Vu TTT, Schneider-Smith E, Aman MJ, Diep BA. Efficacy of Active Immunization With Attenuated alpha-Hemolysin and Panton-Valentine Leukocidin in a Rabbit Model of Staphylococcus aureus Necrotizing Pneumonia. J Infect Dis. 2020 Jan 2;221(2):267-275. doi: 10.1093/infdis/jiz437. PMID 31504652
- [Background] Tree JA, Hall G, Rees P, Vipond J, Funnell SG, Roberts AD. Repeated high-dose (5 x 10(8) TCID50) toxicity study of a third generation smallpox vaccine (IMVAMUNE) in New Zealand white rabbits. Hum Vaccin Immunother. 2016 Jul 2;12(7):1795-801. doi: 10.1080/21645515.2015.1134070. PMID 26836234
- [Background] Tristan A, Ferry T, Durand G, Dauwalder O, Bes M, Lina G, Vandenesch F, Etienne J. Virulence determinants in community and hospital meticillin-resistant Staphylococcus aureus. J Hosp Infect. 2007 Jun;65 Suppl 2:105-9. doi: 10.1016/S0195-6701(07)60025-5. PMID 17540252
- [Background] Venkatasubramaniam A, Adhikari RP, Kort T, Liao GC, Conley S, Abaandou L, Kailasan S, Onodera Y, Krishnan S, Djagbare DM, Holtsberg FW, Karauzum H, Aman MJ. TBA225, a fusion toxoid vaccine for protection and broad neutralization of staphylococcal superantigens. Sci Rep. 2019 Mar 1;9(1):3279. doi: 10.1038/s41598-019-39890-z. PMID 30824769
- [Background] Venkatasubramaniam A, Liao G, Cho E, Adhikari RP, Kort T, Holtsberg FW, Elsass KE, Kobs DJ, Rudge TL Jr, Kauffman KD, Lora NE, Barber DL, Aman MJ, Karauzum H. Safety and Immunogenicity of a 4-Component Toxoid-Based Staphylococcus aureus Vaccine in Rhesus Macaques. Front Immunol. 2021 Feb 25;12:621754. doi: 10.3389/fimmu.2021.621754. eCollection 2021. PMID 33717122
- [Background] Verreault D, Ennis J, Whaley K, Killeen SZ, Karauzum H, Aman MJ, Holtsberg R, Doyle-Meyers L, Didier PJ, Zeitlin L, Roy CJ. Effective Treatment of Staphylococcal Enterotoxin B Aerosol Intoxication in Rhesus Macaques by Using Two Parenterally Administered High-Affinity Monoclonal Antibodies. Antimicrob Agents Chemother. 2019 Apr 25;63(5):e02049-18. doi: 10.1128/AAC.02049-18. Print 2019 May. PMID 30782986
- [Background] Voyich JM, Otto M, Mathema B, Braughton KR, Whitney AR, Welty D, Long RD, Dorward DW, Gardner DJ, Lina G, Kreiswirth BN, DeLeo FR. Is Panton-Valentine leukocidin the major virulence determinant in community-associated methicillin-resistant Staphylococcus aureus disease? J Infect Dis. 2006 Dec 15;194(12):1761-70. doi: 10.1086/509506. Epub 2006 Nov 2. PMID 17109350
- [Background] Wang Y, Mukherjee I, Venkatasubramaniam A, Dikeman D, Orlando N, Zhang J, Ortines R, Mednikov M, Sherchand SP, Kanipakala T, Le T, Shukla S, Ketner M, Adhikari RP, Karauzum H, Aman MJ, Archer NK. Dry and liquid formulations of IBT-V02, a novel multi-component toxoid vaccine, are effective against Staphylococcus aureus isolates from low-to-middle income countries. Front Immunol. 2024 Apr 3;15:1373367. doi: 10.3389/fimmu.2024.1373367. eCollection 2024. PMID 38633244